CLINICAL TRIAL: NCT06619119
Title: Effect of Emergency Escape Room Simulation on Students' Knowledge, Anxiety and Satisfaction Level: Randomized Controlled Study
Brief Title: The Effect of Emergency Escape Room Simulation on Students' Knowledge, Anxiety and Satisfaction Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Hacer Ozel, Assistant Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 01.02.2024/124
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Nursing Education
Keywords: Emergency Nursing; Escape Room; Simulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Escape room simulation group (Experimental): Intervention Group: In addition to the traditional training method within the scope of emergency nursing training, an escape room application was applied to this group after 14 weeks of emergency nursing training.
  Interventions: Other: Excape room simulation
- Control group (No Intervention): Control Group: No intervention other than the traditional education method was applied to this group within the scope of the 14-week emergency nursing education. In the traditional education, narration, question and answer, and discussion techniques were used with a powerpoint presentation containing visuals and text in the classroom environment.

INTERVENTIONS:
Other: Excape room simulation — Application of Research:
  Preparation and Implementation of the Escape Room The escape room game scenario prepared by the relevant faculty members consists of the subjects of Triage, Basic Life Support, Advanced Life Support and Traumas, which are included in the Emergency Nursing course curriculum. Students who will participate in the escape room game were given 30 minutes to solve the puzzles in the room, follow the clues, find the exit key and escape. To solve puzzles, unlock padlocks, and find specific objects in the escape room, students had to answer questions on Triage, Basic Life Support, Advanced Life Support, and Traumas and manage to exit the room in time.
  Arms: Escape room simulation group

SUMMARY:
This research is a randomized controlled study type. The population of the research consisted of a total of 40 students studying at the Hamidiye Nursing Faculty of the University of Health Sciences and taking the emergency nursing course in the 2023-2024 academic year. The sample consisted of nursing students who took this course in the same date range and agreed to participate in the research.

In this study, participants were divided into two equal groups: intervention (n=20) and control group (n=20) using a computer-based randomization method (https://www.random.org/). Due to the nature of the research, the participants and the principal investigator were not blinded, while the evaluator was blinded to the groups.

In addition to the traditional training method within the scope of emergency nursing training, an escape room application was applied to the intervention group after 14 weeks of emergency nursing training.

No intervention other than the traditional education method was applied to the control group within the scope of the 14-week emergency nursing education. In the traditional education, narration, question and answer, and discussion techniques were used in a powerpoint presentation containing visuals and text in the classroom environment.

DETAILED DESCRIPTION:
This research is a randomized controlled study type. The population of the research consisted of a total of 40 students studying at the Hamidiye Nursing Faculty of the University of Health Sciences and taking the emergency nursing course in the 2023-2024 academic year. The sample consisted of nursing students who took this course in the same date range and agreed to participate in the research. In this study, participants were divided into two equal groups: intervention (n=20) and control group (n=20) using a computer-based randomization method (https://www.random.org/). Due to the nature of the research, the participants and the principal investigator were not blinded, while the evaluator was blinded to the groups. In addition to the traditional training method within the scope of emergency nursing training, an escape room application was applied to the intervention group after 14 weeks of emergency nursing training. No intervention other than the traditional training method was applied to the control group within the scope of the 14-week emergency nursing education. Data from the participants were collected through face-to-face interviews using the Personal Information Form, Emergency Nursing Knowledge Test, VAS Satisfaction Scale and State Anxiety Inventory. Participants were informed about the study before the application and filled out a Personal Information Form. Emergency Nursing Knowledge Test, VAS Satisfaction Scale, and State Anxiety Inventory were administered to both groups immediately before and immediately after the escape room simulation application. One week and one month after the application, the Knowledge Test was applied again to both groups. Data collection took approximately 30 minutes. Analysis of data will be performed using IBM SPSS Statistics, version 25.0 (IBM Corporation, Armonk, NY). Descriptive statistical methods such as percentage, mean, standard deviation and median will be used to evaluate the data, and the Kolmogorov-Smirnov distribution test will be used to examine normal distribution. Depending on the characteristics of the variables, chi-square test will be used for categorical data, t-test/Mann Whitney-U test, One-Way ANOVA/Kruskall Wallis tests will be used for measurement data, and Tukey's HSD test/Mann Whitney U test will be used to determine the differences between groups in these tests. Statistical significance will be evaluated at p<0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Being a nursing student
* Having taken the Emergency Nursing course in the 2023-2024 academic year at the Faculty where the research will be conducted

Exclusion Criteria:

* Filling out data collection forms incompletely
* Wanting to leave the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Knowledge level | 5 minutes before and after intervention, 1 week and 1 month after the intervention
  The knowledge test, created by the researchers in line with the literature, consists of 20 questions that question the learning objectives of the Emergency Nursing course and the teaching outcomes of the escape room scenario. Each of the 20 questions asked to the students in the knowledge test was evaluated as 5 points.

SECONDARY OUTCOMES:
Satisfaction level | 5 minutes after intervention
  Visual Analogue Scale (VAS) was used to visualize students' satisfaction with emergency nursing education. Students evaluated themselves on a scale from 1 (very dissatisfied) to 10 (very satisfied) and marked their satisfaction on the visual scale.

OTHER OUTCOMES:
Anxiety level anxiety | 5 minutes before and after intervention
  The anxiety level of the students was measured with the State-Trait Anxiety Inventory.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozel H, Akpinar EG. The Effect of Emergency Escape Room Simulation on Knowledge, Anxiety, and Satisfaction Levels of Students: A Randomized Controlled Trial. Games Health J. 2025 Sep 23. doi: 10.1177/2161783X251378638. Online ahead of print. PMID 40986456